CLINICAL TRIAL: NCT05684029
Title: Near-Infrared Autofluorescence With PTH Test Strip as an SOP of Parathyroid in Thyroid Surgery
Acronym: PTFINDER
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director, Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Other Study IDs: PT FINDER
Record Dates: First submitted 2022-11-27; First posted 2023-01-13 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Cancer; Hypoparathyroidism; Optical Imaging
Keywords: PTH test strip; near-infrared autofluorescence (NIRAF); Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Thyroid surgical specimens, including the thyroid gland, central compartment lymph nodes, and adipose tissue, may include ischemic parathyroid glands. These parathyroid glands, if exist, will transplant back into the patient's body after they are identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Near-infrared Step: 1. Use near-infrared equipment to detect surgical specimens; 2. Timing near-infrared equipment detects parathyroid glands and takes photography; 3. recording the positive tissue in NIRAF; 4. analyzing the accuracy of NIR equipment to see positive points.
  Interventions: Device: Near-infrared devices; Diagnostic Test: PTH test strip
- Senior Surgeon Step: 1. Senior Surgeon inspects for parathyroid glands in postoperative thyroid specimens with the naked eye; 2. Timing senior doctors with parathyroid glands; 3. PTH test strips confirm all suspicious tissues. 4. all analyzing the accuracy of the positive points of senior doctors.
  Interventions: Diagnostic Test: PTH test strip

INTERVENTIONS:
Device: Near-infrared devices — This device can emit and collect near-infrared light of a specific wavelength. The parathyroid glands in the specimen appear as a high-brightness image in the device, to find the parathyroid gland that may be accidentally removed from the specimen.
  Groups: Near-infrared Step
Diagnostic Test: PTH test strip — The PTH test strip is to detect the PTH in the specimen by immunocolloidal gold technology to determine whether it is parathyroid.

SUMMARY:
This is a prospective study aiming to establish near-infrared autofluorescence technology and PTH test strip as a standardized process for finding and identifying parathyroid glands in thyroid surgery.

DETAILED DESCRIPTION:
This is a prospective study aiming to establish near-infrared autofluorescence technology and PTH test strip as a standardized process for finding and identifying parathyroid glands in thyroid surgery.

NIFRA first photographed all specimens from thyroidectomy with or without central neck dissection, and positive tissues under near-infrared light were recorded in a neck map. Then, a senior surgeon examined the parathyroid glands with the naked eye. These suspicious tissues were then identified with the PTH test strip as a gold standard. Finally, the parathyroid glands discovered during the operation that could not be preserved in situ were excluded from the procedure comparison and classified as strategic parathyroid transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with thyroid cancer by FNA
* Scheduled for surgical treatment

Exclusion Criteria:

* Patients with papillary thyroid microcarcinoma who ready for radiofrequency ablation or survival monitoring

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with thyroid cancer by FNA and scheduled for surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Positive tissue identify by NIFRA | During operation, Surgical specimens were photographed with NIRAF, and the location and amount of positive tissue were recorded and marked on the neck map.
  Surgical specimens were photographed with NIRAF, and the location and amount of positive tissue were recorded and marked on the neck map.
Suspicious parathyroid tissue found by surgeons | During operation, Surgeons looked for suspicious parathyroid tissue with the naked eye and These tissues are tested with PTH strips to confirm that they are parathyroid.
  Surgeons looked for suspicious parathyroid tissue with the naked eye and divided them into less than 10% confidence group, 10-90% confidence group, and greater than 90% confidence group. These tissues are tested with PTH strips to confirm that they are parathyroid tissue.
number of strategic parathyroid transplantation | During operation, The parathyroid glands that had been discovered during the operation that could not be preserved in situ were excluded from the procedure comparison and classified as strategic parathyroid transplantation.
  The parathyroid glands that had been discovered during the operation that could not be preserved in situ were excluded from the procedure comparison and classified as strategic parathyroid transplantation.

SECONDARY OUTCOMES:
inspect duration | During operation, From initial examination to finding suspicious parathyroid tissue, excluding subsequent PTH testing steps
  inspect duration in difference method
The number of parathyroid glands in pathological report | Up to 4 weeks, The number of parathyroid glands in pathological report excludes fragments of parathyroid glands less than 3mm in diameter.
  The number of parathyroid glands in pathological report

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No